CLINICAL TRIAL: NCT06037213
Title: Non-interventional Study to Collect Real-world Patient-Reported Outcomes Data in Platinum-Sensitive Relapsed Ovarian Cancer Patients With Long-Term Use of Niraparib
Brief Title: A Real-World Patient-Reported Outcomes Study in Patients With Long-Term Use of Niraparib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-PRO1
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
Keywords: patient-reported outcomes; niraparib; real-world; ovarian cancer; quality of life
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective, non-interventional study is designed to evaluate the quality of life of Chinese ovarian cancer patients with long-term niraparib use in a real-world setting. Participants will complete questionnaires or accept telephone follow-up to provide information about their quality of life.

DETAILED DESCRIPTION:
In this prospective, non-interventional study, patients with platinum-sensitive relapsed ovarian cancer who have received niraparib as maintenance therapy for more than two years will agree to be contacted by questionnaire or telephone three times. The interval will be 4-6 weeks. Information on quality of life will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed platinum-sensitive recurrent epithelial ovarian, fallopian tube or primary peritoneal cancer
* Maintenance treatment with niraparib for ≥2 years and continuing for the next 28 days
* No significant cognitive impairment
* Understand the trial procedure and be able to sign the informed consent form before any study-related procedures

Exclusion Criteria:

* Patients who are not suitable for participation in this study according to the investigator's evaluation
* Patients receiving antineoplastic drugs for other malignancies
* Patients who are unable to comply with the protocol procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Patients are members of the patient assistance programme population.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported health-related quality of life (HRQoL) - EQ-5D-5L questionnaire | 4 months
  The EQ-5D is a standardized measure of health status applicable to a wide range of health conditions and treatments designed by the EuroQoL Group (EQ). It consists of the EQ-5D-5L descriptive system, which comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with each dimension having 5 levels (5L), and the EQ visual analogue scale (EQ VAS)
Patient-reported health-related quality of life (HRQoL) - FOSI questionnaire | 4 months
  The FOSI (Functional Assessment of Cancer Therapy-Ovarian Symptom Index) is a validated tool with eight items that measure response to treatment based on symptom assessment. The questions assess pain, fatigue, nausea, vomiting, bloating, cramping, worry, and QoL. Patients report their symptoms over the past week using a five-point Likert scale, which ranges from 0 (not at all) to 4 (very much).

OTHER OUTCOMES:
Patient population checklist | at baseline
  Baseline characteristics, disease history, comorbidities and concomitant treatments, education.
Niraparib medication checklist | at baseline
  Starting dose, dose modification.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiang, MD., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No